CLINICAL TRIAL: NCT06962098
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Dose-ranging, Multicenter Study to Evaluate the Efficacy and Safety of Isuzinaxib in Subjects With Diabetic Kidney Disease
Brief Title: Efficacy and Safety Study of Isuzinaxib in Subjects With DKD
Acronym: PROMISS-DKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APX-115-05
Record Dates: First submitted 2025-04-16; First posted 2025-05-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: Isuzinaxib; APX-115; NOX; Diabetic Nephropathy; DN; Diabetic Kidney Disease; DKD
MeSH Terms: conditions — Diabetic Nephropathies | interventions — isuzinaxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isuzinaxib 400 mg (Active Comparator): Subject will receive the 400 mg of Isuzinaxib.
  Interventions: Drug: Isuzinaxib
- Isuzinaxib 200 mg (Active Comparator): Subject will receive the 200 mg of Isuzinaxib.
  Interventions: Drug: Isuzinaxib
- Placebo (Placebo Comparator): Subject will receive the Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isuzinaxib — Oral dosing regimen once daily
  Other Names: APX-115
  Arms: Isuzinaxib 200 mg; Isuzinaxib 400 mg
Drug: Placebo — Oral dosing regimen once daily
  Arms: Placebo

SUMMARY:
This study is a multicenter, double-blinded, randomized, placebo-controlled, dose-ranging study to evaluate the safety, tolerability, PK, and efficacy of Isuzinaxib compared with placebo in subjects with DKD.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subject aged ≥19 years inclusive at the time of informed consent.
2. Clinical diagnosis of type 2 diabetes and DKD.
3. 18.5 kg/m² < body mass index < 35 kg/m².
4. Stable UACR values prior to screening visit.
5. UACR between 200 and 3000 mg/g.
6. Hemoglobin A1c ≤10% at Screening Visit.
7. Subject who has been taking unchanged dosage of angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blockers (ARB) medication.
8. Subject who has been on stable anti-hyperglycemic prior to screening.
9. Females of childbearing potential/sexually active males with a partner of childbearing potential: commitment to consistently and correctly use an acceptable method of birth control.
10. Willing to be under dietary management for diabetes.
11. Willing to comply with all study procedures and availability for the duration of the study.
12. Capable of understanding the content of and able voluntarily to provide a signed and dated written informed consent form (ICF) prior to any study procedures.

Exclusion Criteria:

1. History of type 1 diabetes mellitus or gestational diabetes.
2. Subject's renal impairment and/or albuminuria is considered to be of origin other than DKD.
3. History of renal transplant and/or plan to undergo a renal transplant during the study.
4. History of acute kidney injury or renal dialysis.
5. Subject with uncontrolled blood pressure.
6. Subject taking immunosuppressant.
7. Subject with known or suspected hypersensitivity to any components of the APX-115 formulation.
8. Clinically significant abnormal laboratory findings at screening.
9. History of drug or alcohol abuse within 1 year prior to screening.
10. History of any cardiovascular event or cardiovascular procedure planned during the clinical study.
11. Current or history of New York Heart Association class III or IV heart failure.
12. Clinically significant electrocardiogram (ECG) abnormalities.
13. Known significant liver disease.
14. Subject with active urinary tract infection or has not fully recovered before randomization.
15. History of malignancy within 5 years prior to screening.
16. Administration of any investigational product.
17. Major surgery within 28 days or not fully recovered surgery prior to randomization or major surgery planned during the next 6 months.
18. Positive hepatitis B surface antigen.
19. Female subject who is pregnant or breastfeeding.
20. Other medical history which in the opinion of the Investigator would make the subject unsuitable for participation in the study.
21. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study or unable to cooperate because of a language problem or poor mental status.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint: Urine Albumin-Creatinine Ratio | Over 24 Weeks
  Change in Urine Albumin-Creatinine Ratio from baseline through Week 24 in the Isuzinaxib treatment groups versus the placebo group

SECONDARY OUTCOMES:
Efficacy endpoint: eGFR | Over 24 Weeks
  Change from baseline in the eGFR
Efficacy endpoint: Urine Albumin-Creatinine Ratio | Over 20 Weeks
  Change in Urine Albumin-Creatinine Ratio from baseline through Week 20 in the Isuzinaxib treatment groups versus the placebo group
Efficacy endpoint: Urine Albumin-Creatinine Ratio decrease | Over 24 Weeks
  Subjects with a percentage decrease in Urine Albumin-Creatinine Ratio
Efficacy endpoint: Incidence of Composite Renal Outcome | Over 24 Weeks
  Number of subjects with end-stage kidney disease, kidney-related death, or renal replacement therapy
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Over 24 Weeks
  Incidence of treatment-emergent adverse events
PK Endpoint: Pharmacokinetics | Over 24 Weeks
  Assessment of plasma concentrations of Isuzinaxib

OTHER OUTCOMES:
Plasma Biomarkers | Over 24 Weeks
  MCP-1
Urinary Biomarkers | Over 24 Weeks
  KIM-1, NGAL

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Korea University Ansan Hospital, Ansan-si
  - Inje university Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - SoonChunHyang University Hospital Cheonan, Cheonan
  - Keimyung University Daegu Dongsan Hospital, Daegu
  - Inje university Ilsan Paik Hospital, Goyang-si
  - Hanyang University Guri Hospital, Guri-si
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - CHA Bundang Medical Center, Seongnam-si
  - Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdon, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul ST.MARY'S Hospital, Seoul
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan